CLINICAL TRIAL: NCT00622765
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Ranging Study to Investigate the Safety and Efficacy of JNJ-16269110 in Overweight and Obese Subjects
Brief Title: A Study of the Safety and Effectiveness of JNJ-16269110 (R256918) in Overweight and Obese Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR011362; R256918OBE2001
Record Dates: First submitted 2007-12-21; First posted 2008-02-25 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-04

CONDITIONS: Obesity; Nutritional and Metabolic Diseases; Metabolic Diseases; Nutrition Disorders; Overweight
Keywords: Obesity, Overweight, Body Weight, Body Size, Nutritional and Metabolic Diseases
MeSH Terms: conditions — Obesity; Nutritional and Metabolic Diseases; Metabolic Diseases; Nutrition Disorders; Overweight; Body Weight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 001 (Experimental): R256918 5 mg capsule twice daily
  Interventions: Drug: R256918
- 002 (Experimental): R256918 10 mg capsule twice daily
  Interventions: Drug: R256918
- 003 (Experimental): R256918 15 mg capsule twice daily
  Interventions: Drug: R256918
- 004 (Placebo Comparator): placebo Placebo capsule twice daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — Placebo capsule twice daily
  Arms: 004
Drug: R256918 — 5 mg capsule twice daily
  Arms: 001
Drug: R256918 — 10 mg capsule twice daily
  Arms: 002
Drug: R256918 — 15 mg capsule twice daily
  Arms: 003

SUMMARY:
This study investigates the effectiveness and safety of 12 weeks of treatment with JNJ-16269110 (R256918), in overweight and obese patients. The primary measure of effectiveness is the change in body weight at a clinically relevant dosage level during treatment. Additional measures include body mass index (BMI), DEXA (dual X-ray absorptiometry which is a specialized x-ray test that measures body composition), fasting glucose, lipid levels, and blood pressure. Safety assessments performed during the trial include laboratory tests, vital sign measurements, and adverse event reporting.

DETAILED DESCRIPTION:
This is a randomized (assigned study drug by chance), double-blind (both the patient and investigator do not know whether patient is assigned to receive study drug or placebo), placebo-controlled study involving overweight and obese patients. Patients are randomized to one of 4 treatment groups and receive study drug or placebo for a period of 12 weeks. The study consists of 3 phases: a pretreatment phase (including a screening period of 1 week and a period prior to active treatment of 4 weeks), the treatment period of 12 weeks, and a posttreatment phase (consisting of a follow-up visit). Standardized nonpharmacologic therapy (individualized calorie deficit diets containing no more than 30% calories from fat and nutritional counseling) will be administered from Week 4 through the follow-up period. During the treatment period, patients visit the center every two weeks. On each visit, patients come to the clinic after 8 hours fasting. For effectiveness assessments, patients will be weighed and BMI calculated at each visit; waist and hip circumference and DEXA measurements (for body composition and fat mass analysis) will be performed at selected time points. Additional effectiveness assessments from a blood sample include levels of fasting hemoglobin type A1c (HbA1c), glucose, cholesterol, triglycerides, insulin, C-peptide, and gastrointestinal hormones. Insulin sensitivity and pancreas function are evaluated. Safety evaluations, including incidence of adverse events, clinical laboratory results, vital signs, and electrocardiograms, are performed during the study. Patients complete a questionnaire related to stomach/bowel symptoms (GI) throughout the study. Blood samples will also be drawn for an analysis of the subjects genes and an analyses of the body's handling of the study drug. The overall duration of the study for each patient is approximately 19 weeks. The study hypothesis is that treatment with JNJ-16269110 (R256918) will cause a change in body weight compared to placebo and will be well tolerated in overweight and obese patients. This hypothesis will be investigated at each dosage level to determine a clinically relevant dose. 5 mg capsules, 10 mg capsules, 15 mg capsules, or matching placebo capsules taken orally.

ELIGIBILITY:
Inclusion Criteria:

* Obese or overweight at screening defined as: BMI greater than or equal to 30 kg/m2 and <50 kg/m2 or BMI greater than or equal to 27 kg/m2 and <50 kg/m2 in the presence of controlled hypertension and/or treated or untreated dyslipidemia. For patients receiving antihypertensive and/or hypolipidemic medications, these should have been at a stable dosage for at least 2 months before the start of the run-in period. Controlled hypertension is defined as a diastolic blood pressure <100 mmHg and a systolic blood pressure <160 mmHg, in the presence of antihypertensive drug treatment. For patients who are not on lipid-lowering drugs, dyslipidemia is defined as LDL-C greater than or equal to 3.4 mmol/L (130 mg/dL), HDL C <1 mmol/L (40 mg/dL) for men or <1.3 mmol/L (50 mg/dL) for women, or triglycerides greater than or equal to 1.7 mmol/L (150 mg/dL)
* A stable weight, i.e., increasing or decreasing not more than 5 kg in the 3 months before the start of the run-in period
* Consumption of breakfast and dinner on a daily basis
* Ability to swallow the intact capsule (17.5 mm in length and 9.1 mm in diameter) with water, as judged by e.g., the patients's history of having no difficulty with swallowing e.g., capsules or intact tablets
* Fasting plasma glucose <7.0 mmol/L (126 mg/dL) at screening
* Women must be postmenopausal or surgically incapable of childbearing or if sexually active, be practicing an effective method of birth control

Exclusion Criteria:

* History of obesity with a known cause (e.g., Cushing's disease)
* History of anorexia nervosa, bulimia, or binge-eating disorder
* An established diagnosis of diabetes mellitus or treatment with glucose lowering prescription drugs at screening
* Prior exposure or known contraindication or hypersensitivity to R256918
* History of weight-reducing diet or receiving any drugs to treat obesity within the 3 months prior to screening
* Treatment with any investigational drug or device within 1 month before the start of the run-in period
* History or evidence of liver or renal impairment
* History of HIV or presence of hepatitis C antibodies or positive hepatitis B serology
* History of clinically significant gastro-intestinal disease
* History of major gastro-intestinal surgery other than appendectomy or uncomplicated cholecystectomy
* Previous gastric restrictive surgery or other surgical procedures to induce weight loss
* Liposuction within the last 3 months before screening
* Pregnant or nursing women, or women who plan to become pregnant during the study
* History of significant cardiovascular disease or hypertension
* Elevated levels of thyroid-stimulating hormone (TSH)
* A significant change in smoking habits within 3 months of the start of the run-in period
* Malignancy or a history of a malignancy within 5 years before the start of the run-in period, other than basal cell carcinomas of the skin or in situ cervical carcinoma
* History of seizures or significant central nervous system-related disorders
* History of significant psychiatric disorder, including, schizophrenia, or psychosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2007-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Mean change in body weight from baseline to Week 12. | Baseline, 12 weeks

SECONDARY OUTCOMES:
Changes in body weight, body mass index (BMI), body composition, blood pressure, glucose, intestinal hormone levels, beta cell function and lipid parameters. | 12 weeks
Quality of Life scores on questionnaires. | 12 weeks
Safety parameters monitored at each visit. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (18):
- Belgium (2):
  - Edegem
  - Liège
- Denmark (3):
  - Frederiksberg C N/A
  - Hellerup
  - Vipperroed
- Finland (2):
  - Helsinki
  - Kuopio
- Germany (3):
  - Berlin
  - Dresden
  - Heidelberg
- Netherlands (3):
  - Amsterdam
  - Hilversum
  - Rotterdam
- Sweden (2):
  - Gothenburg
  - Huddinge
- United Kingdom (3):
  - Liverpool
  - London
  - Luton

REFERENCES:
- See also: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Dose-Ranging Study to Investigate the Safety and Efficacy of JNJ-16269110 in Overweight and Obese Subjects — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=729&filename=CR011362_CSR.pdf